CLINICAL TRIAL: NCT04999995
Title: To Explore the Potential of UCH-L1 as a Novel Therapeutic and Diagnostic Target in Heart Failure
Brief Title: Diagnostic Potential of UCHL1 in Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CARA-005-19F; 1569386 (Other: William Jennings Bryan Dorn VA Medical Center)
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Dyspnea; Cardiac
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma/serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- HFrEF: Patients admitted with acutely decompensated HFrEF.
- HFpEF: Patients admitted with acutely decompensated HFpEF.
- Non-HF Dyspnea: Patients admitted with acute dyspnea without evidence of HF.

SUMMARY:
Autophagy is considered an important component of Heart failure progression. Deubiquitination enzymes play an important role in autophagy. An important regulatory process within the autophagy pathway is ubiquitination. Ubiquitination targets proteins for degradation. On the contrary, de-ubiquitinating proteins (such as UCHL1) reverses this process. Studies have demonstrated deubiquitination to be linked to certain pathological processes, such as heart failure. UCHL1 will be examined as a potential marker of disease progression in acute decompensated heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is an important cause of morbidity and mortality among US Veterans. Epidemiologic data points to acute decompensated heart failure (ADHF) as a leading cause of hospitalizations in the VA system. The pathophysiologic mechanisms underlying the progressive deterioration of cardiac function remain poorly understood. Autophagy is an evolutionarily conserved pathway that targets cytoplasmic contents to the lysosome for degradation in the cell. In mammals, autophagy has been classified into three different types depending on the means by which the target is delivered into lysosomes for final degradation: (i) macroautophagy, (ii) microautophagy, (iii) chaperone-mediated autophagy (CMA). Both macroautophagy and CMA may participate in degradation of damage proteins; however, only macroautophagy could clear the damage organelles in the cells. Among them, macroautophagy (thereafter and other parts of this proposal referred to as autophagy) is the best characterized. It can be induced by nutrient deprivation and various stress conditions; in these circumstances, autophagy is essential for the maintenance of cell homeostasis by its promotion of the removal of damaged components including long-live and dysfunctional proteins and damaged organelles, such as mitochondria, as well as by its provision of energy and biomolecules to cells including cardiomyocytes. Thus, autophagy is increasingly recognized to play an important role in protecting the heart against various pathological stress-induced damage and dysfunction. In contrast, it has also been proposed that autophagy may be detrimental to the heart in some specific settings. However, the precise reason for such discrepancies is poorly understood. In particularly, the regulatory mechanisms for selective control of autophagy-mediated cardiac protection or dysfunction are unclear. The therapeutic approach targeting autophagy to cardiac disease and heart failure remains to be established.

An important regulatory process within the autophagy pathway is ubiquitination. Ubiquitination targets proteins for degradation. On the contrary, de-ubiquitinating proteins reverses this process. Studies have demonstrated deubiquitination to be linked to certain pathological processes, such as heart failure. Ubiquitin carboxyhydrolase L1 (UCHL1) has been identified by the co-investigator (Dr. Taixing Cui) in mouse models of pressure-overload cardiomyopathy. More data is required to identify UCHL1 as a significant marker in humans with HF.

Heart failure biomarkers play an important role in heart failure care. In general, despite significant overlaps, these biomarkers are loosely arranged into the following categories: 1) myocardial stress/injury, 2) neurohormonal activation, 3) remodeling and 4) comorbidities. None of current biomarkers alone or in combination may fulfil the need regarding screening, diagnosis, prognosis and therapy guidance. Therefore, it is important to find out novel biomarkers of cardiac disease and heart failure, especially those which reflect in important pathophysiologic pathway involved in heart failure disease process and help clinical judgement for understanding diagnosis, prognosis, or management of heart failure. As a result, the novel biomarkers will supplement traditional clinical and laboratory testing to improve understanding of the complex disease processes of heart failure and possibly achieve personalized care for heart failure patients. Human studies of circulating UCHL1 have identified it as a having diagnostic or prognostic value in this pathological settings. However, whether it is applicable to cardiovascular disease has not been studied. This gap will be filled in part by this proposal.

Aim: To explore the diagnostic and/or prognostic value of circulating exosomal UCH-L1 in VA HF patients. We will translate findings from animal models to bed side by a proof-of-principal study to demonstrate that circulating UCH-L1, particularly the exosomal UCH-L1 is higher during acute decompensation than when compensated in VA HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission for decompensated HF (traditional diagnostic criteria will be utilized for diagnosing ADHF - presence of dyspnea as presenting complaint; evidence of volume overload - peripheral or pulmonary edema, elevated jugular venous pressure > 10 cmH2O, presence of hepatojugular reflux, or ascites; elevated B-type Natriuretic Peptide (>100ng/ml); evidence of pulmonary vascular congestion on chest x-ray1, or Admission for dyspnea that is NOT related to ADHF (absence of all HF symptoms and signs mentioned in ADHF inclusion criteria- except for dyspnea as presenting complaint)
* Able to give informed consent
* Age >= 18 years

Exclusion Criteria:

* Mortality during inpatient observation
* Presence of acute stroke (ischemic or hemorrhagic)
* Presence of intracranial hemorrhage
* History of acute stroke (ischemic or hemorrhagic) or intracranial hemorrhage within the preceding 6 months
* Presence of decompensated liver disease (elevated ALT/AST; ascites; Acute variceal bleeding; or hepatic encephalopathy)
* Presence of sepsis
* Presence of severe hyponatremia (Serum sodium < 130 meq/L)
* Active malignancy (undergoing chemotherapy, radiation therapy, or planned surgical intervention)
* SARS-CoV-2 positive during the current admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single Center VA patients with systolic and diastolic HF, acutely decompensated (ADHF), and a comparator cohort with non-HF dyspnea of non-cardiac origin (the control) will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 30 days
  Assess accuracy of UCHL1 to diagnose ADHF as well as correlate with improvement

CONTACTS AND LOCATIONS:
Overall Officials: Taixing Cui, PhD MB, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow VA directives for data sharing.

DOCUMENTS (1):
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04999995/ICF_000.pdf